CLINICAL TRIAL: NCT00732576
Title: Effects of Omega-3 Fatty Acids and Menaquinone-7 on Thrombotic Tendency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Dr. C. Vermeer, VitaK BV
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MEC 07-3-067
Record Dates: First submitted 2007-10-10; First posted 2008-08-12 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2009-03

CONDITIONS: Atherosclerosis
Keywords: Cardiovascular; Calcification
MeSH Terms: conditions — Atherosclerosis; Calcinosis | interventions — menaquinone 7; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 1 (Active Comparator): 9 fish oil capsules, equivalent to 3 gram per day of n-3 polyunsaturated fatty acids (PUFA)
  Interventions: Dietary Supplement: fish oil
- 2 (Active Comparator): 9 fish oil capsules, equivalent to 3 gram per day of n-3 polyunsaturated fatty acids (PUFA) including 1 capsule of menaquinone-7 per day (10 µg)
  Interventions: Dietary Supplement: menaquinone-7; Dietary Supplement: fish oil
- 3 (Active Comparator): 9 fish oil capsules, equivalent to 3 gram per day of n-3 polyunsaturated fatty acids (PUFA) including 2 capsules of menaquinone-7 per day (20 µg per day)
  Interventions: Dietary Supplement: menaquinone-7; Dietary Supplement: fish oil
- 4 (Active Comparator): 9 fish oil capsules, equivalent to 3 gram per day of n-3 polyunsaturated fatty acids (PUFA) including 1 capsule of menaquinone-7 per day (45 µg per day)
  Interventions: Dietary Supplement: menaquinone-7; Dietary Supplement: fish oil
- 5 (Active Comparator): 9 krill oil capsules, equivalent to 1,5 gram per day of n-3 polyunsaturated fatty acids (PUFA)
  Interventions: Dietary Supplement: krill oil
- 6 (Active Comparator): 9 krill oil capsules, equivalent to 1,5 gram per day of n-3 polyunsaturated fatty acids (PUFA) including 1 capsule of menaquinone-7 per day (10 µg)
  Interventions: Dietary Supplement: menaquinone-7; Dietary Supplement: krill oil
- 7 (Active Comparator): 9 krill oil capsules, equivalent to 1,5 gram per day of n-3 polyunsaturated fatty acids (PUFA) including 2 capsules of menaquinone-7 per day (20 µg per day)
  Interventions: Dietary Supplement: menaquinone-7; Dietary Supplement: krill oil
- 8 (Active Comparator): 9 krill oil capsules, equivalent to 1,5 gram per day of n-3 polyunsaturated fatty acids (PUFA) including 1 capsule of menaquinone-7 per day (45 µg per day)
  Interventions: Dietary Supplement: menaquinone-7; Dietary Supplement: krill oil

INTERVENTIONS:
Dietary Supplement: menaquinone-7 — capsule consisting of 10, 20 or 45 µg menaquinone-7 per day during 8 weeks
  Other Names: MenaQ7
  Arms: 2; 3; 4; 6; 7; 8
Dietary Supplement: fish oil — 9 fish oil capsules equivalent to 3 gram per day of n-3 polyunsaturated fatty acids during 12 weeks
  Arms: 1; 2; 3; 4
Dietary Supplement: krill oil — 9 krill oil capsules, equivalent to 1,5 gram per day of n-3 polyunsaturated fatty acids (PUFA) during 12 weeks
  Arms: 5; 6; 7; 8

SUMMARY:
Omega-3 fatty acids are notably present in fish oil and krill oil, and are known to have beneficial effects on the vasculature. Vitamin K2 is known for preventing vascular calcification. In this study we investigate a potential synergy between the effects of either fish or krill oil and menaquinone-7, which is one of K2 vitamins.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects - BMI < 30
* written informed consent

Exclusion Criteria:

* Use of oral anticoagulants
* Coagulation disorders
* Use of multivitamin supplements
* Use of corticosteroids, anticonceptives
* hypertriglyceridemia, hypercholesterolemia

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Endogenous Thrombin Potential (ETP) | 12 weeks

SECONDARY OUTCOMES:
Osteocalcin carboxylation | 12 weeks
Matrix Gla-protein carboxylation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — Department of Biochemistry, Maastricht University
Locations (1):
- VitaK - Maastricht University, Maastricht, Netherlands